CLINICAL TRIAL: NCT02190955
Title: Assessment of the Educational Experience for Patients With Newly Diagnosed Nephrotic Syndrome
Brief Title: Assessment of the Educational Experiences for Patients Newly Diagnosed With Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Maine Medical Partners (Unknown); C.S. Mott Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 6802
Record Dates: First submitted 2014-05-30; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NEPTUNE contact registry patients: Patients and caregivers will be recruited from the Nephrotic Syndrome Study Network (NEPTUNE) Patient Contact Registry. Over 1000 patients and caregivers are members of the registry and have already provided permission to be contacted for future research studies. Analysis of the one-time online questionnaire will be done in collaboration with investigators from the NEPTUNE Consortium.

SUMMARY:
The purpose of this study is to learn about patient, caregiver and healthcare worker perspectives on educating patients with newly-diagnosed Nephrotic Syndrome. All patients enrolled in the Contact Registry with Nephrotic Syndrome will be invited via email to participate in this study.

DETAILED DESCRIPTION:
The survey included questions addressing the following areas: 1.) Information that is important to know when learning to manage Nephrotic Syndrome. 2.) Preferred resources for the education of patients and caregivers with newly-diagnosed Nephrotic Syndrome. 3.) The time frame required to acquire confidence in the management of Nephrotic Syndrome. 4.) Disease-specific information such as diagnosis, length of disease duration, medications used, need for kidney biopsy, dialysis and/or transplant. 5.) Demographic data such as race/ethnicity and educational background.

The survey data is stored by the Rare Diseases Clinical Research Network's Data Management and Coordinating Center (DMCC) at the University of South Florida. The data is de-identified. Names or other personal health information were not collected. Upon conclusion of the study period, the data will be sent to the NEPTUNE consortium lead at the University of Michigan.

ELIGIBILITY:
Inclusion Criteria:

Patient and Patient Caregiver:

* 18 years or older
* English literate
* History of Nephrotic Syndrome > 3 months or caregiver of a child diagnosed with Nephrotic Syndrome > 3 months prior to enrollment
* Informed Consent

Healthcare Worker Inclusion Criteria:

* Age > 18 years
* English literate
* Provides medical care for children or adults with Nephrotic Syndrome
* Informed Consent

Exclusion Criteria:

* Inability to provide informed consent and complete survey
* Other criteria as specified by Consortium and based on the data we collect in the Contact Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and caregivers were recruited from the Nephrotic Syndrome Study Network (NEPTUNE) Patient Contact Registry. Over 1000 patients and caregivers are members of the registry and have already provided permission to be contacted for future research studies. The Contact Registry was created to inform patients and/or parents of patients with Nephrotic Syndrome of clinical research studies.
  Health professionals, including pediatric and internal medicine nephrologists and nephrology nurses will be recruited from the 18 NEPTUNE study network sites.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Stakeholder perspectives about educational experiences of newly-diagnosed Nephrotic Syndrome patients | 1 year after the study is closed to enrollment
  The outcome measure(s) will be evaluated based on the cross-sectional online questionnaire. The questionnaire is the only study procedure for this online patient contact registry protocol and will be the sole analysis tool for both the primary and secondary outcome measures.

SECONDARY OUTCOMES:
Perspectives of patients/families with healthcare workers regarding educational needs of newly-diagnosed Nephrotic Syndrome | 1 year after the study is closed to enrollment
  The outcome measure(s) will be evaluated based on the cross-sectional online questionnaire. The questionnaire is the only study procedure for this online patient contact registry protocol and will be the sole analysis tool for both the primary and secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Tanzer, MD, Study Chair — Maine Medical Partners; Debbie Gipson, MD, Study Chair — C.S. Mott Children's Hospital
Locations (1):
- University of South Florida Data Management and Coordinating Center, Tampa, Florida, United States